CLINICAL TRIAL: NCT00495521
Title: A Prospective Randomized Double-Blind Study of PASER® in the Management of Patients Experiencing an Acute Flare of Crohn's Disease
Brief Title: High Dose Oral 4-Aminosalicylic Acid (PASER®) to Control Acute Flares of Mild to Moderate Crohn's Disease in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efforts at recruitment have halted as recruitment was poor
Sponsor: Jacobus Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PASER - AFC.002
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's; Crohn's Disease; Acute Flare; Mild to Moderate Crohn's Disease; Children; Pediatrics; Ileo-cecal; Pediatric Crohn's Disease; New Onset Crohn's Disease; Recently diagnosed Crohn's Disease
MeSH Terms: conditions — Crohn Disease; Pediatric Crohn's disease | interventions — Aminosalicylic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): 4-Aminosalicylic acid extended release granules (as volume equivalent of active product), 50 mg/kg orally three times daily for two weeks followed by (as volume equivalent) 50 mg/kg orally two times daily for 2 weeks
  Interventions: Drug: 4-Aminosalicylic acid extended release granules
- Placebo (Placebo Comparator): Placebo granules identical in appearance to the active arm (as volume equivalent of active product), 0 mg/kg orally three times daily for two weeks followed by (as volume equivalent) 0 mg/kg orally two times daily for 2 weeks
  Interventions: Drug: 4-Aminosalicylic acid extended release granules

INTERVENTIONS:
Drug: 4-Aminosalicylic acid extended release granules — Granules for oral administration will be administered as a volume equivalent to 50 mg/kg of 4-aminosalicylic acid three times daily for 2 weeks followed by 2 times daily for 2 weeks in the active arm or a comparable volume in the placebo arm
  Other Names: PASER® Granules (or Placebo Granules); 4-Aminosalicylic acid; NDC 49938-107-04; 4-ASA

SUMMARY:
The purpose of this 4 week study is to determine whether PASER®, an approved delayed-release oral formulation of 4-aminosalicylic acid, in doses of 50 milligrams per kilogram three times daily for 2 weeks followed by 50 milligrams per kilogram twice daily for 2 weeks, will resolve an acute flare of ileocecal Crohn's disease.

DETAILED DESCRIPTION:
Eligible pediatric patients with acute flares of ileocecal Crohn's disease will be randomized to receive either PASER®, an approved delayed-release oral formulation of 4-aminosalicylic acid, in doses of 50 milligrams per kilogram three times daily for 2 weeks followed by 50 milligrams per kilogram twice daily for 2 weeks, or an identical-appearing placebo preparation.

Patients will be required to maintain a daily diary and to return at 2 weeks for blood and stool tests. At the four week mark, patients will return for clinical evaluation, global assessment of disease activity and change in disease activity, as well as additional laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 18 years
* Crohn's disease predominantly involving the ileum and/or cecum. The diagnosis must have been established by radiography, endoscopy and/or biopsy (at least 2 of the 3 modalities) with at least one confirmatory test having been performed no more than 36 months before entry. The diagnosis must have been confirmed by at least one gastroenterologist.
* Harvey Bradshaw Index of at least 7
* The onset of the acute flare should have been abrupt, declaring itself over 72 hours, and should have started no more than 4 weeks before study entry. Symptoms relating to the flare should not have diminished or started to improve prior to entry.
* Written informed consent

Exclusion Criteria:

* Concomitant corticosteroids, budesonide
* Corticosteroids within 2 months
* Cyclosporine, mycophenolate mofetil or experimental drugs during the last three months
* Maintenance infliximab, or infliximab or other biologics in the preceding 3 months
* If the severity of the flare has started to decrease spontaneously
* Coexisting diagnosis of primary sclerosing cholangitis
* Infectious diarrhea
* Signs of intestinal obstruction or perforation
* New fistulization as part of the acute flare or increased activity in chronic fistula(e) as part of the acute flare
* Hypersensitivity to 4-ASA or any components of PASER®
* Pregnancy or breast-feeding
* Failure of a woman of child-bearing potential to agree to use adequate contraception for the 4 week period of the trial, if sexually active
* Severe renal or hepatic disease (i.e., more than 3 times upper limit of normal) or a WBC < 3,000 during the preceding three months

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Jacobus, MD, Study Chair — Jacobus Pharmaceutical; Kathy L Ales, MD, Study Director — Jacobus Pharmaceutical; George D Ferry, MD, Principal Investigator — Texas Children's Hospital, Baylor College of Medicine; Marla C Dubinsky, MD, Principal Investigator — Cedars-Sinai Medical Center; Joel R Rosh, MD, Principal Investigator — Atlantic Health System, Morristown General Hospital, Goryeb Children's Hospital; Melvin B. Heyman, M.D., M.P.H., Principal Investigator — University of California, San Francisco; Stanley A. Cohen, M.D., Principal Investigator — Children's Center for Digestive Healthcare, LLC
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Children's Center for Digestive HealthCare, LLC, Atlanta, Georgia
  - Atlantic Health System / Morristown Memorial Hospital / Goryeb Children's Hospital, Morristown, New Jersey
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to eligible patients under the care of or referred to investigators at 5 different academic medical centers from July 2007 through October 2008.
Pre-assignment Details: Recruitment was slow with only 2 patients entered.
Groups:
- Active: Oral granules administered as (volume equivalent of active product) 50 mg/kg three times daily for two weeks followed by (volume equivalent) 50 mg/kg two times daily for 2 weeks
- Placebo: Oral granules administered as (volume equivalent of active product) 0 mg/kg three times daily for two weeks followed by (volume equivalent) 0 mg/kg two times daily for 2 weeks
Period: Overall Study
Arm/Group | Active | Placebo
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 4-Aminosalicylic Acid Extended Release Granules: Oral granules administered as (volume equivalent of active product) 50 mg/kg three times daily for two weeks followed by (volume equivalent) 50 mg/kg two times daily for 2 weeks
- Placebo Granules: Oral granules administered as (volume equivalent of active product) 0 mg/kg three times daily for two weeks followed by (volume equivalent) 0 mg/kg two times daily for 2 weeks
- Total: Total of all reporting groups
Arm/Group | 4-Aminosalicylic Acid Extended Release Granules | Placebo Granules | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 12 [12 to 12] | 14 [14 to 14] | 13 [12 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Reduction in the Modified Crohn's Disease Activity Index (mCDAI) Score of >70 Points by 4 Weeks Compared With Baseline
Description: Reduction in the Modified Crohn's Disease Activity Index (mCDAI) score of >70 points by 4 weeks after randomization compared with baseline
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 1 | 1
participants | 1 | 1

2. Secondary Outcome: Rate of Remission
Description: Rate of remission was defined by a decrease in modified Crohn's Disease Activity Index (mCDAI) > 100 points and total mCDAI < 150 by 4 weeks
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

3. Secondary Outcome: Rate of Response as Defined by a Reduction in HBI to Less Than 5 by 4 Weeks
Time Frame: 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Rate of Remission as Defined by the Decrease in HBI to Less Than 3 by 4 Weeks
Time Frame: 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Response and/or Remission Including Time to Change in HBI, According to Elements of the Daily Patient Diary
Time Frame: up to 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Rate of Response as Defined by the Decrease in PCDAI of 12.5 Points by 4 Weeks
Time Frame: 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Rate of Remission as Defined by the Decrease in PCDAI < 10 by 4 Weeks
Time Frame: 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in IMPACT-III From Baseline to 4 Weeks
Time Frame: 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in the Patient's General Sense of Disease Activity as Recorded in the Individual Daily Diary
Time Frame: 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Absence of Night Time Stools, if They Were Present on Entry, and Time to Disappearance
Time Frame: up to 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Normalization of All Other Components in the Diary
Time Frame: up to 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Hgb, ESR, CRP, Platelet Count, Calprotectin From Baseline and Time to Normalization
Time Frame: 2 weeks and 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Global Physician Assessment of Disease Activity From Baseline to Study Completion
Time Frame: 4 weeks
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of treatment
Groups:
- Placebo: Oral granules administered as (volume equivalent of active product) 50 mg/kg three times daily for two weeks followed by (volume equivalent) 50 mg/kg two times daily for 2 weeks
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=1) | Placebo (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Probably related, resolved with change in vehicle of administration and decreased dose
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) — Unlikey to be related; resolved
Worsening of disease, abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Occurred after the 4 week trial during continued off-study use
Chest pain and headache (General disorders) | 0 (0) | 1 (1) — Related to introduction of flaxseed oil and resolved with discontinuation of flaxseed oil
Dizziness after exercise (General disorders) | 0 (0) | 1 (1) — Occurred twice

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No